CLINICAL TRIAL: NCT02066506
Title: Study of Adaptation of the Right Ventricle to Systemic Afterload
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P080609
Record Dates: First submitted 2013-09-17; First posted 2014-02-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2012-08

CONDITIONS: Congenital Heart Disease With Systemic Right Ventricle
Keywords: systemic right ventricle; cardiac magnetic resonance imaging; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- asymptomatic group (Sham Comparator): patients with systemic right ventricle who are asymptomatic,
  Interventions: Other: asymptomatic group
- symptomatic group (Sham Comparator): symptomatic group : patients with systemic right ventricle and heart failure signs and/or decrease exercise performance
  Interventions: Other: symptomatic group
- control (Sham Comparator): healthy subject matched with patients of asymptomatic group
  Interventions: Other: asymptomatic group; Other: symptomatic group

INTERVENTIONS:
Other: asymptomatic group — 2 visits with MRI
  Arms: asymptomatic group; control
Other: symptomatic group — 2 visits with MRI
  Arms: control; symptomatic group

SUMMARY:
the first purpose of the study is to determine the adaptative mechanisms of right ventricle (RV) to systemic afterload, and the mechanisms of RV failure, in patients with congenital heart disease and subaortic RV, using cardiac magnetic resonance imaging (CMR).The mechanisms are evaluated by measures of RV remodelling and RV wall stress using CMR. Second objectives are to evaluate these mechanisms using echography, arterial properties study and neurohormonal levels

DETAILED DESCRIPTION:
Right ventricle (RV) in sub-aortic position is a rare situation, mainly in two congenital heart defects: congenitally corrected transposition of the great arteries and complete transposition of the great arteries palliated by atrial switch. In these patients, increase of afterload leads to hypertrophy and late RV dilatation. The stress exercised on RV walls could play a role in adaptative mechanisms to systemic afterload. Beyond a remodelling threshold, it could cause fibrosis damage and RV systolic failure. Magnetic resonance imaging, which has a major potential in estimation of RV remodelling, wall stress and fibrosis, could shed light on RV adaptation to systemic afterload and evolution towards failure. Systemic RV remodelling and function could also depend on the neuro-hormone secretion and mechanical arterial properties, that have a direct influence on patients afterload. The first purpose of the study is to determine the adaptative mechanisms of RV to systemic afterload, and the mechanisms of RV failure, in patients with congenital heart disease and subaortic RV, using cardiac magnetic resonance imaging (CMR).The mechanisms are evaluated by measures of RV remodelling and RV wall stress using CMR. Second objectives are to evaluate these mechanisms using echography, arterial properties study and neurohormonal levels

ELIGIBILITY:
Patients inclusion criteria:

* patients with a systemic right ventricle
* to have an insurance
* to obtain informed consent

Patients non-inclusion criteria:

* patients with cyanosis defined by a saturation ≤ 85% at rest
* patients with a ventricular septal defect non repaired at the time of inclusion
* contraindications normal MRI
* contraindication to achieving a stress test
* Glomerular Filtration Rate inf 30ml/mn/1.73m²
* physical or mental disability that does not allow to perform a cardiopulmonary exercise test
* patients with already severe allergy to gadolinium MRI contrast
* current Pregnancy
* patients who can not be monitored over the period of one year, patient participating in another research on the Treatment interacting with the neurohormonal system in particular the renin-angiotensin-aldosterone system

healthy subjects inclusion criteria:

* matched for age and sex + / - 5 years of an asymptomatic patient
* Normal ECG
* normal Echocardiography
* clinical examination prior
* Patient receiving an insurance
* Obtaining informed consent

healthy subjects Exclusion criteria:

* History of myocardial infarction-known or detectable on the ECG-abnormal Liver function tests
* Complete Blood Count
* electrolytes
* viral serology
* Primary or secondary cardiomyopathy-known or detectable on echocardiography
* History of thoracic radiotherapy or chemotherapy
* Contraindications MRI
* Counter-indication for performing a stress test
* Patient with severe renal clearance less than Glomerular Filtration Rate inf 30ml/mn/1.73m²
* Patient has already made a severe allergy to gadolinium MRI contrast Current Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
remodelling indexes | 48 months
wall stress index | 48 months
fibrosis of systemic RV measured by MRI | 48 months

SECONDARY OUTCOMES:
echographic measures of RV function and geometry indexes | 48 months
  comparison between patients and healthy subjects and analysis of the evolution of the measured parameters in the 2 groups after one year of follow
Arterial mechanical properties (stiffness aortic distensibility and arterial compliance) | 48 months
  comparison between patients and healthy subjects and analysis of the evolution of the measured parameters in the 2 groups after one year of follow
Rate of neurohormones of the renin-angiotensin-aldosterone system and neuropeptides | 48 months
Variability and reproducibility indices remodeling and wall stress MRI | 48 months
  inter and intra-observer variability and inter-examination MRI measures

CONTACTS AND LOCATIONS:
Overall Officials: Magalie Ladouceur, MD, Principal Investigator — Université Paris Descartes
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France